CLINICAL TRIAL: NCT02782078
Title: Pharmacological Interaction of Rifampicin on Clindamycin in Staphylococcic Osteoarticular Infections
Acronym: DALARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140318 / AOR14027
Record Dates: First submitted 2016-05-02; First posted 2016-05-25 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Staphylococcal Infections
Keywords: osteoarticular infection; rifampicin; clindamycin; enzymatic induction; antibiotherapy resistance
MeSH Terms: conditions — Staphylococcal Infections | interventions — Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clindamycin and rifampicin dosages (Other): blood samples for clindamycin and rifampicin dosages (for each patient)
  Interventions: Biological: Clindamycin and rifampicin dosages

INTERVENTIONS:
Biological: Clindamycin and rifampicin dosages — blood samples for clindamycin and rifampicin dosages (for each patient)

SUMMARY:
Clindamycin and rifampicin are authorized in osteoarticular infection treatment (IDSA guidelines) but some interaction is observed. The objective of this study is to evaluate and quantify rifampicin interaction on clindamycin

DETAILED DESCRIPTION:
It could suggest modification of recommended doses or incitement to antibiotic dosage. Thus, theses antibiotics, if association is allowed, could limit fluoroquinolones prescription and avoid some antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥18 years of age
* osteoarticular infection
* staphylococcus detected in bacteriological sampling
* sensibility to rifampicin, erythromycin and clindamycin
* active intravenous antibiotherapy against staphylococcus detected in bacteriological sampling

Exclusion Criteria:

* septic shock or severe initial sepsis
* osteoarticular infection with other microorganism than staphylococcus
* contraindication to clindamycin or rifampicin including case of hypersensibility to one of these two antibiotics
* pre-existing renal insufficiency or severe renal insufficiency (creatinine clearance <30 ml/min)
* serious cognitive disorders
* patient under guardianship, trusteeship or non affiliated to social security or CMU (beneficiary or assignee)
* refusal to take part in the study and to sign the consent form
* pregnancy
* lactation
* administration of clindamycin or rifampicin within the month before inclusion
* treatment with enzymatic inductor or inhibitor within the month before inclusion
* participation to another study modifying antibiotic treatment administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
clindamycin AUC (area under curve) at steady state and after rifampicin introduction | clindamycin AUC will be evaluated after rifampicin interaction, so at day 14 of introduction
  this AUC of clindamycin will be compared to AUC before rifampicin introduction, at day 0

SECONDARY OUTCOMES:
rifampicin auto induction | AUC of rifampicin at day 4 (before autoinduction ant at steady state) and day 14 (after autoinduction)
  rifampicin autoinduction will be studied with rifampicin AUC, according time, for each patient, at day 4 and day 14. Comparison of AUC with student's test
clinical outcome | at day 4, day 14, day 28 (or day 60 if osteosynthesis)
  resolution of symptoms first described (pain, swelling, fever…) with specific scale
biological outcome | at day 4, day 14, day 28 (or day 60 if osteosynthesis)
  resolution of inflammatory syndrome (measure of C reactive protein) and hyperleucocytosis (WBC)
side effects and toxicity: number of participants with treatment related adverse events as assessed by CTCAE v4.0 | at day 2, day 4, day 14, day 28 (or day 60 if osteosynthesis)
  skin lesion, digestive symptoms, clostridium infection, liver cytolysis, hematological disorders (leucopenia, hemolytic anemia, thrombopenia)…

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine Goulenok, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Interne - Hôpital Bichat Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No